CLINICAL TRIAL: NCT05928429
Title: Effects of Cryotherapy on Objective and Subjective Symptoms of Taxane-Induced Neuropathy in Patients With Early Breast Cancer: A National, Multicenter, Prospective, Randomized, Controlled Trial
Brief Title: Effects of Cryotherapy on Taxane-Induced Neuropathy in Patients With Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Lendorf (Other)
Collaborators: Danish Cancer Society (Other); Aarhus University Hospital (Other); Nordsjaellands Hospital (Other); Hospital of Southern Jutland (Other)
Responsible Party: Sponsor-Investigator, Maria Lendorf, MD, PhD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CryoPac
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: CIPN - Chemotherapy-Induced Peripheral Neuropathy; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: A national, multicenter, interventional, randomized, non-blinded clinical trial evaluating the preventive effects of cryotherapy for CIPN.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm A - interventional (Experimental): Each patient in the experimental arm will wear glycerine-containing Elasto-Gel™ gloves and socks (Elasto-Gel™ mitts for hands: TM7008, and slippers for feet: SL3000; Southwest Technologies, Inc., North Kansas City, MO, USA) over a disposable glove and sock liner secured by Velcro at the wrist and ankle on their hands and feet from 15 minutes before paclitaxel administration to 15 minutes after the infusion is complete (90 minutes in total).
  Interventions: Device: Elasto-Gel™ mitts for hands: TM7008, and slippers for feet: SL3000; Southwest Technologies, Inc., North Kansas City, MO, USA
- arm B (No Intervention): Patients will receive planned paclitaxel chemotherapy without cryotherapy intervention.

INTERVENTIONS:
Device: Elasto-Gel™ mitts for hands: TM7008, and slippers for feet: SL3000; Southwest Technologies, Inc., North Kansas City, MO, USA — Patients in the experimental arm will wear glycerine-containing Elasto-Gel™ gloves and socks (Elasto-Gel™ mitts for hands: TM7008, and slippers for feet: SL3000; Southwest Technologies, Inc., North Kansas City, MO, USA) over a disposable glove and sock liner secured by Velcro at the wrist and ankle on their hands and feet from 15 minutes before paclitaxel administration to 15 minutes after the infusion is complete (90 minutes in total).
  Arms: arm A - interventional

SUMMARY:
Due to well-proven survival benefit, paclitaxel and other taxane-based chemotherapies are first-line agents for both the adjuvant and neoadjuvant treatment of early stage breast cancer. Chemotherapy-induced peripheral neuropathy (CIPN) is a frequent and disabling side effect of taxane anticancer agents. No established strategy exists for CIPN prevention. This study is designed to assess the efficacy and safety of cryotherapy for the prevention of paclitaxel-induced peripheral neuropathy in patients with breast cancer in a prospective randomized controlled trial.

DETAILED DESCRIPTION:
BACKGROUND: Due to well-proven survival benefit, paclitaxel and other taxane-based chemotherapies are first-line agents for both the adjuvant and neoadjuvant treatment of early stage breast cancer. Chemotherapy-induced peripheral neuropathy (CIPN) is a frequent and disabling side effect of taxane anticancer agents. No established strategy exists for CIPN prevention. This study is designed to assess the efficacy and safety of cryotherapy for the prevention of paclitaxel-induced peripheral neuropathy in patients with breast cancer in a prospective randomized controlled trial.

OBJECTIVES:

Primary objective: To assess the efficacy of cryotherapy to prevent paclitaxel chemotherapy induced peripheral neuropathy (CIPN) Secondary objective: To search for risk factors for CIPN. METHOD Study Design: A national, multicenter, interventional, randomized, non-blinded clinical trial evaluating the preventive effects of cryotherapy for CIPN.

Eligibility: Key inclusion criteria; Patients with early breast cancer scheduled to receive weekly paclitaxel (80mg/m2 for one hour) 9 doses, PS 0-1.

Sample size: 300 Randomization: Participants will be randomized 1:1 to A: use of Elasto-Gel™ frozen glove and sock on their hands and feet during paclitaxel treatment or B: standard treatment. Randomization will be performed in REDCap using the Electronic Case Report Forms (eCRFs).

Cryotherapy Intervention: Patients in the experimental arm will wear glycerine-containing Elasto-Gel™ gloves and socks (Elasto-Gel™ mitts for hands: TM7008, and slippers for feet: SL3000; Southwest Technologies, Inc., North Kansas City, MO, USA) over a disposable glove and sock liner secured by Velcro at the wrist and ankle on their hands and feet from 15 minutes before paclitaxel administration to 15 minutes after the infusion is complete (90 minutes in total).

Primary outcomes: Incidence of peripheral neuropathy; CIPN is assessed using the Total Neuropathy Score reduced version (TNSr) 21 days after last completed cycle of paclitaxel and compared to baseline.

Key secondary outcomes: Objective symptoms - Quantitative sensory testing (QST).

Subjective symptoms - Patient Reported Outcome: (EORTC Quality of Life Questionnaire (QLQ)-C30 and EORTC (QLQ)-CIPN20), pain and tolerability etc.

ELIGIBILITY:
Inclusion Criteria:

Key inclusion criteria; Patients with early breast cancer scheduled to receive weekly paclitaxel (80mg/m2 for one hour) 9 or 12 doses, PS 0-1

Exclusion Criteria:

Peripheral sensory/motor neuropathy, neuralgia or edema of the limb graded >=2 (CTCAE ver 5.0), Patient with Raynaud's symptoms; peripheral arterial ischemia; or any other reasons based on the primary physician's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of peripheral neuropathy | CIPN is assessed 21 days after last completed cycle of paclitaxel and compared to baseline.
  CIPN is assessed using the Total Neuropathy Score reduced version (TNSr)

CONTACTS AND LOCATIONS:
Locations (1):
- Maria E Lendorf, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No